CLINICAL TRIAL: NCT02830178
Title: Channeling in the Use of Nonprescription Paracetamol and Ibuprofen in an Electronic Medical Records Database: Evidence and Implications
Brief Title: A Study of Channeling in the Use of Nonprescription Paracetamol and Ibuprofen in an Electronic Medical Records Database: Evidence and Implications
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RRA-16387; RRA-16387 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-06-07; First posted 2016-07-12 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Hemorrhage, Gastrointestinal; Myocardial Infarction; Stroke; Kidney Diseases
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Myocardial Infarction; Stroke; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Any Paracetamol: Participants with age 18 and over who received a first prescription of single-ingredient paracetamol or ibuprofen in 2012 will be enrolled. Their status with respect to prior gastrointestinal bleeding, myocardial infarction, stroke, or kidney disease will be assessed based on the presence or absence of a diagnosis in the 2 years prior to the index date. This observational study will evaluate whether new users of paracetamol have a higher prevalence of certain conditions (gastrointestinal bleeding, myocardial infarction, stroke or kidney disease) in their history when compared to new users of ibuprofen, propensity scores and outcome models.
- Ibuprofen: Participants with age 18 and over who received a first prescription of single-ingredient ibuprofen in 2012 will be enrolled. Their status with respect to prior gastrointestinal bleeding, myocardial infarction, stroke, or kidney disease will be assessed based on the presence or absence of a diagnosis in the 2 years prior to the index date. This observational study will evaluate whether new users of paracetamol have a higher prevalence of certain conditions (gastrointestinal bleeding, myocardial infarction, stroke or kidney disease) in their history when compared to new users of ibuprofen, propensity scores and outcome models.

SUMMARY:
The Purpose of this study is to examine whether evidence of channeling exists by analyzing within a cohort of participants with first prescriptions of single-ingredient paracetamol or ibuprofen (or both) whether participants with paracetamol were more likely to have an ibuprofen-related contraindication.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in up-to-standard practices (practices that have been qualified for research purposes by the Clinical Practice Research Datalink [CPRD] administrators) in the CPRD
* Received a first prescription for paracetamol or a first prescription for ibuprofen in 2012
* Were age 18 or older in the date of their qualifying prescription in 2012

Exclusion Criteria:

* Who received a prescription for paracetamol or ibuprofen in the 6 months prior to their qualifying prescription in 2012
* Who received a prescription for any acetaminophen- or ibuprofen-containing combination products in the 6 months prior to the qualifying prescription in 2012

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is a cohort of participants 18 and over who received a first prescription of single-ingredient paracetamol or ibuprofen in 2012.
Sampling Method: Non-Probability Sample
Enrollment: 144337 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evidence of Channeling as Measured by an Odds-ratio Different From 1.0 for Contraindications to Ibuprofen Comparing Paracetamol and Ibuprofen Groups | up to 7 months
  Participants receiving first prescriptions of single-ingredient paracetamol or ibuprofen will be assessed to analyze whether participants with paracetamol were more likely to have had an ibuprofen-related contraindication than participants with ibuprofen.

SECONDARY OUTCOMES:
Propensity Score Model | up to 7 months
  The potential to control for channeling bias will be examined. It will also assess whether there will be sufficient overlap in propensity scores to allow for adequate adjustment to control for bias due to channeling. The propensity score is the estimated probability of receiving a treatment (paracetamol), based on the available data, ranges from 0 to 1. The higher the score, the more likely to be treated with paracetamol.
Extent of Bias as Measured by an Odds-ratio Different From 1.0 for the Covariate Indicating Exposure to Paracetamol or Ibuprofen in the Negative Control Outcome Models | up to 7 months
  Relative risks for paracetamol versus ibuprofen for the 31 negative control outcomes should be 1.0 if there is no bias. A series of models with increasing numbers of covariates will be fit to measure the extent to which covariates can diminish the impact of bias.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Raritan, New Jersey, United States

REFERENCES:
- [Derived] Weinstein RB, Ryan P, Berlin JA, Matcho A, Schuemie M, Swerdel J, Patel K, Fife D. Channeling in the Use of Nonprescription Paracetamol and Ibuprofen in an Electronic Medical Records Database: Evidence and Implications. Drug Saf. 2017 Dec;40(12):1279-1292. doi: 10.1007/s40264-017-0581-7. PMID 28780741